CLINICAL TRIAL: NCT02334722
Title: A Shortened Antiepileptic Drug (AED) Course in Surgical Brain Tumor Patients: A Randomized Trial
Brief Title: 1 Week Versus 6 Weeks of Levetiracetam in Surgical Brain Tumor Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201400876; OCR14673 (Other: University of Florida)
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Results first posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Brain Neoplasms; Brain Cancer; Brain Tumors; Cancer of the Brain; Cancer of Brain; Seizure
MeSH Terms: conditions — Brain Neoplasms; Seizures | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 Week Levetiracetam (Experimental): Levetiracetam taken by mouth at a daily dose of 1000 mg for one week.
  Interventions: Drug: Levetiracetam
- 6 Week Levetiracetam (Active Comparator): Levetiracetam taken by mouth at a daily dose of 1000 mg for six weeks.
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam
  Other Names: Keppra

SUMMARY:
The purpose of this study is to see if there are any differences in patient reported neurotoxicity between patients who receive Levetiracetam tablets for one week after surgery to remove a brain tumor versus those who receive Levetiracetam tablets for six weeks after surgery. Specifically, we will see if one group has less side effects than the other, and whether or not one group has more seizures than the other.

DETAILED DESCRIPTION:
Because seizures are one of the leading neurologic complications in brain tumor patients, neurosurgeons prescribe antiepileptic drugs (AEDs) to help prevent them. Although the American Academy of Neurology (AAN) guidelines recommend that AEDs be stopped after the first post-operative week in patients without seizures, there is no standard length of treatment and some patients may stay on AEDs indefinitely.

In an attempt to develop clinical guidelines for AED use in post-operative brain tumor patients, we will try to determine if taking levetiracetam for 1 week results in less neurotoxicity than taking it for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years of age and older) patients who have or will have undergone surgical resection or biopsy of a supratentorial brain tumor and are able to consent for themselves.
* Able to be randomized prior to or up to 48 hours after surgery.

Exclusion Criteria:

* No known history of seizure activity.
* Pregnant or breastfeeding.
* Renal dysfunction (CrCl < 30ml/min).
* Beck's Depression Inventory (BDI) ≥14
* Allergy to levetiracetam.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-08-05 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Rahman, MS, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled in this trial on 8/5/2015 and the last on 8/27/2020 at an academic medical center in a Neurosurgical inpatient/outpatient setting. Potential participants were adult (>18 years of age and older) patients, with no seizure history, who had or will have had undergone surgical resection of a supratentorial brain tumor and were able to consent for themselves.
Groups:
- 1 Week Levetiracetam: Levetiracetam taken by mouth at a daily dose of 1000 mg for one week.
  Levetiracetam
- 6 Week Levetiracetam: Levetiracetam taken by mouth at a daily dose of 1000 mg for six weeks.
  Levetiracetam
Period: Overall Study
Arm/Group | 1 Week Levetiracetam | 6 Week Levetiracetam
Started | 40 | 41
Completed | 33 | 34
Not Completed | 7 | 7
Not completed — Lost to Follow-up | 4 | 0
Not completed — 6 week questionnaire not completed | 2 | 0
Not completed — Unable to obtain medication | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Subjects were screened against eligibility criteria. Subjects with a history of seizures, depression or use of psychiatric medications, Beck-Depression Inventory score over 14, biopsy only or other factors were determined ineligible. Potential participants who may have been eligible also declined participation.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Week Levetiracetam | 6 Week Levetiracetam | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age of participants in each arm
  years | 59.8 (13.7) | 49.9 (17.1) | 54.8 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Percent of subjects that are male or female.
  Participants
    Female | 22 | 17 | 39
    Male | 18 | 24 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Percentage of participants identifying as a particular ethnicity in each arm
  Participants
    Hispanic or Latino | 2 | 2 | 4
    Not Hispanic or Latino | 37 | 39 | 76
    Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Percentage of participants identifying as a particular race in each arm
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 3 | 5
    White | 37 | 38 | 75
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 40 | 41 | 81

OUTCOME MEASURES:

1. Primary Outcome: Change in Neurotoxicity Scale Scores
Description: The Neurotoxicity Scale is as a validated 27 question, patient-reported measure for assessing the adverse effects of antiepileptic drugs on cognitive function. Patients self-report "no problem", "a mild problem", "a moderate problem" or "a serious problem" for each question corresponding to a score of 0, 1, 2, and 3, respectively. For each patient, the overall score was formed by summing scores in all 27 questions. The minimum possible score is 0 and the maximum possible total score is 81. A lower score indicates less toxicity when taking an antiepileptic drug. The outcome is a score change from baseline at the 6 week follow-up and is calculated by subtracting the baseline score from the 6 week follow-up score for each patient.
Time Frame: Baseline to 6 weeks
Population: All patients taking levetiracetam 1000 mg daily, not stratified by dosing schedule.
Measure: Median (Full Range); unit: score on scale
Arm/Group | 1 Week Levetiracetam | 6 Week Levetiracetam
Number analyzed (Participants) | 33 | 34
score on scale | -1 [-22 to 38] | -3.5 [-18 to 38]
Statistical Analysis 1: Comparison: 1 Week Levetiracetam vs 6 Week Levetiracetam; Test type: Superiority; p = 0.7824, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -2.5

ADVERSE EVENTS:
Time Frame: Adverse events will be collected from first dose of study drug to six week evaluation or sooner if the patient contacts their physician/study team about new symptoms/problems.
Description: Participants at risk for all-cause mortality included any participant who signed consent to take part in the study. Participants at risk for Serious Adverse Events and Other (not including serious) Adverse Events included only participants who received study intervention.
Arm/Group | 1 Week Levetiracetam | 6 Week Levetiracetam
All-Cause Mortality (participants affected / at risk) | 2/40 | 0/41
Serious Adverse Events (participants affected / at risk) | 11/39 | 7/37
Other Adverse Events (participants affected / at risk) | 27/39 | 22/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Week Levetiracetam (N=39) | 6 Week Levetiracetam (N=37)
Aphasia (Nervous system disorders) | 3 (3) | 0 (0)
Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cerebral edema (Nervous system disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 3 (3) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Weakness (Nervous system disorders) | 0 (0) | 1 (1)
Pseudomeningocele (Nervous system disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Spinal Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 0 (0)
Hip Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mental Status Change (Nervous system disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Week Levetiracetam (N=39) | 6 Week Levetiracetam (N=37)
Fatigue (General disorders) | 6 (7) | 8 (9)
Headache (Nervous system disorders) | 9 (9) | 6 (6)
Confusion (Nervous system disorders) | 3 (4) | 5 (6)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 4 (4)
Nausea (Gastrointestinal disorders) | 7 (7) | 5 (5)
Aphasia (Nervous system disorders) | 2 (2) | 2 (2)
Facial Swelling (Gastrointestinal disorders) | 3 (3) | 2 (2)
Incision Pain (General disorders) | 3 (3) | 3 (3)
Mental Status Change (Psychiatric disorders) | 4 (4) | 3 (3)
Seizure (Nervous system disorders) | 2 (2) | 2 (3)
Vision Change (Eye disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/22/NCT02334722/Prot_SAP_000.pdf